CLINICAL TRIAL: NCT05186116
Title: Living Donor Liver Transplantation (LDLT) in Non Resectable Colo-rectal Cancer Liver Metastasis. The LIVERMORE Trial (LIVing Donor livEr tRansplant Modena cOloRectal mEtastasis) [Original Title in Italian: "Trapianto di Fegato da Donatore Vivente Per Metastasi Epatiche Non Resecabili da Adenocarcinoma Del Colon"]
Brief Title: LDLT in Non Resectable Colo-rectal Cancer Liver Metastasis
Acronym: LIVERMORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Fabrizio Di Benedetto, Professor, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 470/2021/SPER/AOUMO
Record Dates: First submitted 2021-11-24; First posted 2022-01-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Colon Adenocarcinoma; Liver Metastasis Colon Cancer
Keywords: LDLT; living donor; CRLM; transplant oncology
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LDLT, partial graft, whole graft recipients (Experimental): Patients that undergo LDLT, partial graft or whole graft transplantation for CRLM in the study period
  Interventions: Procedure: Living donor liver transplant, Split liver transplant, RAPID, DDLT

INTERVENTIONS:
Procedure: Living donor liver transplant, Split liver transplant, RAPID, DDLT — Transplantation of part of the liver from a living donor, or entire cadaveric graft

SUMMARY:
This study is an interventional open label prospective study that aims to assess both overall and disease-free survival of patients treated with LDLT, partial or whole graft LT from deceased donors for unresectable CRLM.

Secondary outcomes are graft survival and donor outcomes in terms of safety and quality of life.

Donor selection is performed according to the currently used Institutional and National standards and protocols.

DETAILED DESCRIPTION:
Liver Transplant (LT) is a feasible, safe and effective curative strategy for patients with unresectable colorectal liver metastases (CRLM), and several trials are currently active and in a recruitment phase to study its impact with both conventional donors and living donors (LDLT).

As a matter of fact, in this setting living donors represent a helpful resource, thanks to the opportunity to schedule the LT at the timeliest conditions in terms of oncological response and patient's performance status. LDLT is a well-established procedure that is already offered to patients listed for LT at our Institution.

Crucial requirement for study eligibility is the assessment of non-resectability of the presented liver metastases from colorectal cancer (CRC).

Criteria for non-resectability of the liver-only CRC metastases eligible for the study should be assessed at the patient study entry, by the surgeon in charge together with the multidisciplinary team.

Patients fulfilling the inclusion criteria of the study will undergo clinical, translational and regulatory steps. Briefly, the main procedures and requirements of the study can be summarized as follows:

- Pre-transplant screening and waiting phase:

Screening of patients with liver-limited CRC metastases potentially eligible to the study will be registered. The screening for general eligibility to liver transplantation will be conducted according to the existing Institutional protocol (called in Italian "PDTA", "Percorso Diagnostico Terapeutico Assistenziale").

During screening or waiting time periods, patients will continue planned chemotherapy treatment and will undergo blood tests (including CEA and Ca19.9), thoraco-abdominal CT scan and positron emission tomography (PET) scan (if needed) every 8 weeks.

- Donors' screening:

Screening of donors will be held according to the existing Institutional protocol for LDLT

- Informed consent:

Consent to the study will be signed after completion of the pre-LT screening, that is once co-morbidities and transplant eligibility will be ascertained on top of cancer conditions. In addition, patients will have to sign additional written informed consent prior to any study procedure.

- Post-transplant follow-up:

Following LDLT, standard institutional follow-up procedures will be performed and registered. Patient/graft condition and tumor status should be re-assessed at least every 4 months for the first 3 years, every 6 months for the rest of follow-up.

Following donation standard institutional follow up will be performed on donors and registered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18.
* Histologically confirmed colon and rectum (intraperitoneal) adenocarcinoma.
* Pathological classification of primary tumor as pT1-3, without peritoneal tumor deposits, absence of mucinous component >50%, confirmed R0 resection, no limitations for RAS mutations, B-RAF wild type.
* No signs of extra hepatic metastatic disease or local recurrence according to CT scan+MRI+PET/CT scans.
* Liver metastases not eligible for curative liver resection
* Objective response according to RECIST 1.1 to first-line treatment, with sustained response for at least 4 months, OR disease control (complete [CR] or partial response [PR] or standard disease [SD]) during second- line treatment for at least 4 months.
* Carcinoembryonic Antigen (CEA) values stable or decreasing during the enrollment prior to liver transplant.
* Performance status, ECOG (Eastern Cooperative Oncology Group) 0-2.
* Signed informed consent and expected cooperation of the patients for the treatment and follow-up, and national/local regulations.

Exclusion Criteria:

* Hereditary CRC syndromes including FAP (Familial adenomatous polyposis) and Lynch syndrome.
* Prior extra hepatic metastatic disease or primary tumor local relapse.
* Palliative resection of primary CRC tumor.
* Disease progression
* Other malignancies in the previous 5 years (with exception of in situ cervical carcinoma and basal cell carcinoma; superficial bladder tumors are allowed if curatively treated).
* Active intra-venous or alcohol abusers (patients may be eligible if abstention > 6 months is demonstrated)
* Active HIV infection
* Psychiatric disorders and patient low compliance
* Any reason why, in the judgment of the investigators, the patient should not participate (to be formally declared)

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival of patients treated with LDLT for unresectable CRLM compared to our historical cohort of potentially transplantable patients that underwent chemotherapy only
Disease free survival | 5 years
  Disease-free survival of patients treated with LDLT for unresectable CRLM compared to our historical cohort of potentially transplantable patients that underwent chemotherapy only

SECONDARY OUTCOMES:
Graft survival | 5 years
  Incidence of retransplant in the LDLT group
Donor quality of life | 5 years
  Measure of Health-related quality of life (HRQOL) of donors using the a Short Form Health Survey 36 (SF-36). SF-36 is a multiplanar scale with scores ranging from 0 to 100 where zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Modena, Modena, MO, Italy

REFERENCES:
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Fong Y, Fortner J, Sun RL, Brennan MF, Blumgart LH. Clinical score for predicting recurrence after hepatic resection for metastatic colorectal cancer: analysis of 1001 consecutive cases. Ann Surg. 1999 Sep;230(3):309-18; discussion 318-21. doi: 10.1097/00000658-199909000-00004. PMID 10493478
- [Background] Abdalla EK, Hicks ME, Vauthey JN. Portal vein embolization: rationale, technique and future prospects. Br J Surg. 2001 Feb;88(2):165-75. doi: 10.1046/j.1365-2168.2001.01658.x. PMID 11167863
- [Background] Cremolini C, Casagrande M, Loupakis F, Aprile G, Bergamo F, Masi G, Moretto R R, Pietrantonio F, Marmorino F, Zucchelli G, Tomasello G, Tonini G, Allegrini G, Granetto C, Ferrari L, Urbani L, Cillo U, Pilati P, Sensi E, Pellegrinelli A, Milione M, Fontanini G, Falcone A. Efficacy of FOLFOXIRI plus bevacizumab in liver-limited metastatic colorectal cancer: A pooled analysis of clinical studies by Gruppo Oncologico del Nord Ovest. Eur J Cancer. 2017 Mar;73:74-84. doi: 10.1016/j.ejca.2016.10.028. Epub 2016 Dec 13. PMID 27986363
- [Background] Lang H, de Santibanes E, Schlitt HJ, Malago M, van Gulik T, Machado MA, Jovine E, Heinrich S, Ettorre GM, Chan A, Hernandez-Alejandro R, Robles Campos R, Sandstrom P, Linecker M, Clavien PA. 10th Anniversary of ALPPS-Lessons Learned and quo Vadis. Ann Surg. 2019 Jan;269(1):114-119. doi: 10.1097/SLA.0000000000002797. PMID 29727331
- [Background] Wicherts DA, de Haas RJ, Salloum C, Andreani P, Pascal G, Sotirov D, Adam R, Castaing D, Azoulay D. Repeat hepatectomy for recurrent colorectal metastases. Br J Surg. 2013 May;100(6):808-18. doi: 10.1002/bjs.9088. Epub 2013 Mar 12. PMID 23494765
- [Background] Butte JM, Gonen M, Allen PJ, Peter Kingham T, Sofocleous CT, DeMatteo RP, Fong Y, Kemeny NE, Jarnagin WR, D'Angelica MI. Recurrence After Partial Hepatectomy for Metastatic Colorectal Cancer: Potentially Curative Role of Salvage Repeat Resection. Ann Surg Oncol. 2015 Aug;22(8):2761-71. doi: 10.1245/s10434-015-4370-1. Epub 2015 Jan 9. PMID 25572686
- [Background] Kanas GP, Taylor A, Primrose JN, Langeberg WJ, Kelsh MA, Mowat FS, Alexander DD, Choti MA, Poston G. Survival after liver resection in metastatic colorectal cancer: review and meta-analysis of prognostic factors. Clin Epidemiol. 2012;4:283-301. doi: 10.2147/CLEP.S34285. Epub 2012 Nov 7. PMID 23152705
- [Background] Pawlik TM, Schulick RD, Choti MA. Expanding criteria for resectability of colorectal liver metastases. Oncologist. 2008 Jan;13(1):51-64. doi: 10.1634/theoncologist.2007-0142. PMID 18245012
- [Background] Tsai MS, Su YH, Ho MC, Liang JT, Chen TP, Lai HS, Lee PH. Clinicopathological features and prognosis in resectable synchronous and metachronous colorectal liver metastasis. Ann Surg Oncol. 2007 Feb;14(2):786-94. doi: 10.1245/s10434-006-9215-5. Epub 2006 Nov 14. PMID 17103254
- [Background] Hill CR, Chagpar RB, Callender GG, Brown RE, Gilbert JE, Martin RC 2nd, McMasters KM, Scoggins CR. recurrence following hepatectomy for metastatic colorectal cancer: development of a model that predicts patterns of recurrence and survival. Ann Surg Oncol. 2012 Jan;19(1):139-44. doi: 10.1245/s10434-011-1921-y. Epub 2011 Jul 13. PMID 21751045
- [Background] Muhlbacher F, Huk I, Steininger R, Gnant M, Gotzinger P, Wamser P, Banhegyi C, Piza F. Is orthotopic liver transplantation a feasible treatment for secondary cancer of the liver? Transplant Proc. 1991 Feb;23(1 Pt 2):1567-8. No abstract available. PMID 1989293
- [Background] Toso C, Pinto Marques H, Andres A, Castro Sousa F, Adam R, Kalil A, Clavien PA, Furtado E, Barroso E, Bismuth H; Compagnons Hepato-Biliaires Group. Liver transplantation for colorectal liver metastasis: Survival without recurrence can be achieved. Liver Transpl. 2017 Aug;23(8):1073-1076. doi: 10.1002/lt.24791. No abstract available. PMID 28544246
- [Background] Grut H, Dueland S, Line PD, Revheim ME. The prognostic value of 18F-FDG PET/CT prior to liver transplantation for nonresectable colorectal liver metastases. Eur J Nucl Med Mol Imaging. 2018 Feb;45(2):218-225. doi: 10.1007/s00259-017-3843-9. Epub 2017 Oct 12. PMID 29026950
- [Background] D'Angelica M, Kornprat P, Gonen M, DeMatteo RP, Fong Y, Blumgart LH, Jarnagin WR. Effect on outcome of recurrence patterns after hepatectomy for colorectal metastases. Ann Surg Oncol. 2011 Apr;18(4):1096-103. doi: 10.1245/s10434-010-1409-1. Epub 2010 Nov 2. PMID 21042942
- [Background] Moris D, Tsilimigras DI, Chakedis J, Beal EW, Felekouras E, Vernadakis S, Schizas D, Fung JJ, Pawlik TM. Liver transplantation for unresectable colorectal liver metastases: A systematic review. J Surg Oncol. 2017 Sep;116(3):288-297. doi: 10.1002/jso.24671. Epub 2017 May 17. PMID 28513862
- [Background] Hagness M, Foss A, Egge TS, Dueland S. Patterns of recurrence after liver transplantation for nonresectable liver metastases from colorectal cancer. Ann Surg Oncol. 2014 Apr;21(4):1323-9. doi: 10.1245/s10434-013-3449-9. Epub 2013 Dec 27. PMID 24370906
- [Background] Dueland S, Syversveen T, Solheim JM, Solberg S, Grut H, Bjornbeth BA, Hagness M, Line PD. Survival Following Liver Transplantation for Patients With Nonresectable Liver-only Colorectal Metastases. Ann Surg. 2020 Feb;271(2):212-218. doi: 10.1097/SLA.0000000000003404. PMID 31188200
- [Background] Grut H, Solberg S, Seierstad T, Revheim ME, Egge TS, Larsen SG, Line PD, Dueland S. Growth rates of pulmonary metastases after liver transplantation for unresectable colorectal liver metastases. Br J Surg. 2018 Feb;105(3):295-301. doi: 10.1002/bjs.10651. Epub 2017 Nov 23. PMID 29168565
- [Background] Line PD, Hagness M, Berstad AE, Foss A, Dueland S. A Novel Concept for Partial Liver Transplantation in Nonresectable Colorectal Liver Metastases: The RAPID Concept. Ann Surg. 2015 Jul;262(1):e5-9. doi: 10.1097/SLA.0000000000001165. PMID 25692361
- [Background] Konigsrainer A, Templin S, Capobianco I, Konigsrainer I, Bitzer M, Zender L, Sipos B, Kanz L, Wagner S, Nadalin S. Paradigm Shift in the Management of Irresectable Colorectal Liver Metastases: Living Donor Auxiliary Partial Orthotopic Liver Transplantation in Combination With Two-stage Hepatectomy (LD-RAPID). Ann Surg. 2019 Aug;270(2):327-332. doi: 10.1097/SLA.0000000000002861. PMID 29916882
- [Background] Grat M, Krawczyk M, Stypulkowski J, Morawski M, Krasnodebski M, Wasilewicz M, Lewandowski Z, Grat K, Patkowski W, Zieniewicz K. Prognostic Relevance of a Complete Pathologic Response in Liver Transplantation for Hepatocellular Carcinoma. Ann Surg Oncol. 2019 Dec;26(13):4556-4565. doi: 10.1245/s10434-019-07811-z. Epub 2019 Sep 13. PMID 31520204
- [Background] Dueland S, Foss A, Solheim JM, Hagness M, Line PD. Survival following liver transplantation for liver-only colorectal metastases compared with hepatocellular carcinoma. Br J Surg. 2018 May;105(6):736-742. doi: 10.1002/bjs.10769. Epub 2018 Mar 13. PMID 29532908
- [Background] Dueland S, Grut H, Syversveen T, Hagness M, Line PD. Selection criteria related to long-term survival following liver transplantation for colorectal liver metastasis. Am J Transplant. 2020 Feb;20(2):530-537. doi: 10.1111/ajt.15682. Epub 2019 Nov 28. PMID 31674105
- [Background] Missiaglia E, Jacobs B, D'Ario G, Di Narzo AF, Soneson C, Budinska E, Popovici V, Vecchione L, Gerster S, Yan P, Roth AD, Klingbiel D, Bosman FT, Delorenzi M, Tejpar S. Distal and proximal colon cancers differ in terms of molecular, pathological, and clinical features. Ann Oncol. 2014 Oct;25(10):1995-2001. doi: 10.1093/annonc/mdu275. Epub 2014 Jul 23. PMID 25057166
- [Background] Brudvik KW, Vauthey JN. Surgery: KRAS mutations and hepatic recurrence after treatment of colorectal liver metastases. Nat Rev Gastroenterol Hepatol. 2017 Nov;14(11):638-639. doi: 10.1038/nrgastro.2017.129. Epub 2017 Sep 20. No abstract available. PMID 28930294
- [Background] Marcus L, Lemery SJ, Keegan P, Pazdur R. FDA Approval Summary: Pembrolizumab for the Treatment of Microsatellite Instability-High Solid Tumors. Clin Cancer Res. 2019 Jul 1;25(13):3753-3758. doi: 10.1158/1078-0432.CCR-18-4070. Epub 2019 Feb 20. PMID 30787022
- [Background] Sartore-Bianchi A, Trusolino L, Martino C, Bencardino K, Lonardi S, Bergamo F, Zagonel V, Leone F, Depetris I, Martinelli E, Troiani T, Ciardiello F, Racca P, Bertotti A, Siravegna G, Torri V, Amatu A, Ghezzi S, Marrapese G, Palmeri L, Valtorta E, Cassingena A, Lauricella C, Vanzulli A, Regge D, Veronese S, Comoglio PM, Bardelli A, Marsoni S, Siena S. Dual-targeted therapy with trastuzumab and lapatinib in treatment-refractory, KRAS codon 12/13 wild-type, HER2-positive metastatic colorectal cancer (HERACLES): a proof-of-concept, multicentre, open-label, phase 2 trial. Lancet Oncol. 2016 Jun;17(6):738-746. doi: 10.1016/S1470-2045(16)00150-9. Epub 2016 Apr 20. PMID 27108243
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Line PD, Ruffolo LI, Toso C, Dueland S, Nadalin S, Hernandez-Alejandro R. Liver transplantation for colorectal liver metastases: What do we need to know? Int J Surg. 2020 Oct;82S:87-92. doi: 10.1016/j.ijsu.2020.03.079. Epub 2020 Apr 17. PMID 32305529
- [Background] Sinha PK, Mohapatra N, Bharathy KG, Kumar G, Pamecha V. A Long-Term Prospective Study of Quality of Life, Abdominal Symptoms, and Cosmesis of Donors After Hepatectomy for Live-Donor Liver Transplantation. J Clin Exp Hepatol. 2021 Sep-Oct;11(5):579-585. doi: 10.1016/j.jceh.2020.11.005. Epub 2020 Dec 7. PMID 34511819
- [Background] Bonney GK, Chew CA, Lodge P, Hubbard J, Halazun KJ, Trunecka P, Muiesan P, Mirza DF, Isaac J, Laing RW, Iyer SG, Chee CE, Yong WP, Muthiah MD, Panaro F, Sanabria J, Grothey A, Moodley K, Chau I, Chan ACY, Wang CC, Menon K, Sapisochin G, Hagness M, Dueland S, Line PD, Adam R. Liver transplantation for non-resectable colorectal liver metastases: the International Hepato-Pancreato-Biliary Association consensus guidelines. Lancet Gastroenterol Hepatol. 2021 Nov;6(11):933-946. doi: 10.1016/S2468-1253(21)00219-3. Epub 2021 Sep 8. PMID 34506756
- [Background] Ladner DP, Dew MA, Forney S, Gillespie BW, Brown RS Jr, Merion RM, Freise CE, Hayashi PH, Hong JC, Ashworth A, Berg CL, Burton JR Jr, Shaked A, Butt Z. Long-term quality of life after liver donation in the adult to adult living donor liver transplantation cohort study (A2ALL). J Hepatol. 2015 Feb;62(2):346-53. doi: 10.1016/j.jhep.2014.08.043. Epub 2014 Sep 6. PMID 25195558